CLINICAL TRIAL: NCT03084562
Title: Descriptive Study Comparing Regadenoson Versus Dipyridamole in Use as Pharmacological Stress Agent Before a Myocardial Perfusion Imaging by Single Photon Emission Computed Tomography (SPECT)
Brief Title: Regadenoson vs Dipyridamole in Use as Pharmacological Stress Agent Before SPECT
Acronym: REDUCE
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0056
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2017-03

CONDITIONS: Myocardial Perfusion Imaging
MeSH Terms: interventions — Functional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dipyridamole: stress test impossible or contraindicated (first intention)
  Interventions: Other: collect examination time, functional and clinical tolerability
- Regadenoson: stress test and dipyridamole impossible or contraindicated. In particular, patients with severe COPD or asthmatic patient. (second intention)
  Interventions: Other: collect examination time, functional and clinical tolerability

INTERVENTIONS:
Other: collect examination time, functional and clinical tolerability — Examination time : time from patient setup and launch of the pre-test to the end of the patient monitoring Functional tolerability : functional assessed by the patient Clinical tolerability : clinical score by the cardiologist

SUMMARY:
Myocardial perfusion scintigraphy is to evaluate coronary perfusion as well as heart muscle function. This examination takes place in two stages, one imaging at rest and one after a cardiac stress caused. This stress can be triggered as a first-line stress test. A pharmacological stress is proposed when stress test is not possible or contraindicated, Several drugs have a marketing authorization in this indication (adenosine, dipyridamole, regadenoson, dobutamine).

Among them, the regadenoson is the most recent molecule. Marketed in France since 2013, it would allow a reduction of undesirable effects compared to other agents, especially adenosine. It is simple and quick to use thanks to a single dose administration. However, its cost is nearly 30 times higher than dipyridamole. In the investigational center, dipyridamole is currently the first-line pharmacological stress agent, whereas regadenoson is reserved for a limited number of doses, the indication of which must be justified (asthmatic patient or with severe COPD). Few studies in the literature specifically compare these two pharmacological agents (examination time, cost, tolerance) and the opinion on the use of regadenoson in the service is limited.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Myocardial scintigraphy by pharmacological stress agent
* Used molecules = Dipyridamole or Regadenoson

Exclusion Criteria:

* Physical stress test by single or mixed effort (associating pharmacological stress)
* Pharmacological agent used = Adenosine
* Inclusion in the ERCAD protocol
* Double isotope protocol
* Patient refusal due to study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reffered for an indication of myocardial perfusion scintigraphy in the nuclear medicine unit
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
Duration of the test | 24 hours (Visit 1: During the examen)
  Evaluate the time savings from the use of regadenoson versus dipyridamole by comparing the duration of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Christian SCHEIBER, Pr, Principal Investigator — Lyon civil Hospital - Est Hospital Complexe - Nuclear Medicine Service
Locations (1):
- Lyon civil Hospital - Est Hospital Complexe - Nuclear Medicine Service, Bron, France